CLINICAL TRIAL: NCT00473798
Title: Patient Satisfaction and Psychological Distress Related to Emerging Technologies for Cervical Cancer Screening and Diagnosis
Brief Title: Patient Satisfaction & Quality Of Life in Patients With Cervical Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BS98-269
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Psychosocial; Cervical Cancer
Keywords: Patient Satisfaction; Quality of Life; Psychological Distress; Cervical Cancer; Cervical Cancer Screening; Questionnaire
MeSH Terms: conditions — Uterine Cervical Neoplasms; Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- A: Women who are eligible to participate in a study of the technical feasibility of optical spectroscopy will be invited to participate in this study.
  Interventions: Behavioral: Questionnaire
- A': Women who are eligible to participate in a study of the technical feasibility of optical spectroscopy will be invited to participate in this study.
  Interventions: Behavioral: Questionnaire
- B: Patients who have consented to participate in a randomized trial of optical spectroscopy.
  Interventions: Behavioral: Questionnaire
- C: Women who are eligible to participate in a study of the technical feasibility of optical spectroscopy will be invited to participate in this study.
  Interventions: Behavioral: Questionnaire
- D: Health care providers.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire

SUMMARY:
Primary Objectives:

1. To compare levels of patient anxiety, pain, and satisfaction associated with optical spectroscopy procedures and MDC with the levels associated with colposcopically-directed biopsy in the cervical cancer diagnostic setting and with Papanicolaou smear in the screening setting. This aim will be addressed in Studies A and A' -- Procedure-Related Distress and Patient Satisfaction.
2. To evaluate differences in psychological distress, satisfaction, and adherence to treatment in the two arms of a randomized trial; one group will be diagnosed with usual care procedures (Papanicolaou smear and colposcopically-directed biopsy) plus optical spectroscopy and the second will receive usual care. Aim 2 will be accomplished in Study B -- Psychological Distress, Satisfaction, and Adherence Outcomes in a Randomized Trial of Optical Spectroscopy.
3. To assess the psychosocial and behavioral impact of a false positive screening result. This will be done in Study C -- Impact of False Positive Screening Test on Psychological Distress and Future Screening Intentions.
4. To assess provider receptivity to optical spectroscopy. Aim 4 will be accomplished in Study D -- Survey of Health Care Providers.

DETAILED DESCRIPTION:
Randomized Clinical Trial:

Participants in this study will be interviewed before and after they see the doctor for their first visit. They will be asked about their moods and the tests used to detect cervical cancer. They will also be asked about their symptom, how it is affecting their lives, and their satisfaction with their visit.

Participants will be called approximately 2 weeks, 6 weeks, and 3 months after their appointments to answer questions about their health and quality of life, and the test and treatment they received. In addition, the participants will complete assessments at the 6, 12, 18, and 24 month clinic visits. If participants do not return for these follow-up appointments, the research staff will attempt to contact the participants to do brief interview by phone.

Research staff will also review participant's medical records and gather information on diagnosis, treatment plans and adherence.

This is an investigational study. A total of 360 patients will take part in this multicenter study. About 180 participants at M. D. Anderson will take part in this study.

Studies A and A Prime:

Participants in this study will be interviewed before they see the doctor. They will be asked about their moods and the tests used to detect cervical cancer.

During the medical tests, participants will rate their pain and how tense they are. Someone will watch them to see whether they are upset or in pain. After they see the doctor, participants will be interviewed again about their mood and how much they liked or did not like the test.

Some participants will be interviewed about their opinion of the test at the appointment when they receive their test results. Some participants will complete the Sequelae of LEEP/biopsy and medication use questionnaire. Some participants will be called 7 to 14 days and/or three months after their appointments. Some participants may answer some of the questions on a computer as well as in an interview. They will be asked to answer questions about their moods and about getting tests to detect cervical cancer. A sample of the participants will be selected to have their results visit tape recorded and to answer a few questions about what the doctor told them.

Participants may be contacted to participate in discussion groups about tests for cervical dysplasia. Participation in the discussion groups is voluntary. Research staff will also review participant's medical records and gather information on diagnosis, treatment plans and adherence.

This is an investigational study. A total of 3980 patients will take part in this multicenter study. About 2400 participants at M. D. Anderson will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Studies A, A', and pilot tests

   * Eligible to participate in Project 2
   * Over 18
   * Referred for an abnormal pap or has no history of abnormal pap
   * Consented to participate in the patient outcomes project.
2. Study B

   * Consented to participate in Project 3
   * Over 18
   * Referred for an abnormal pap
   * Consented to participate in the patient outcome project.
3. Study C

   * Same as Study B.
4. Study D

   * Members of the American Society for Colposcopy and Cervical Pathology (ASCCP).

Exclusion Criteria:

1. Studies A, A', and pilot tests through C:

   * Pregnancy
   * Unable to communicate in English, Spanish, or Chinese
2. Study D

   * None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are eligible to participate in a study of the technical feasibility of optical spectroscopy. Total Accrual for Study A: 3510; Study A': 350; pilot tests for Study A': 120; Study B: 360; and Study C: 645. Health care providers will participate in Study D with a total accrual of 900.
Sampling Method: Probability Sample
Enrollment: 1938 (Actual)
Dates: Start 1999-07-01 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Compare levels of patient anxiety, pain, and satisfaction associated with optical spectroscopy procedures and MDC with the levels associated with colposcopically-directed biopsy | 9 Years
Evaluate differences in psychological distress, satisfaction, and adherence to treatment. | 9 Years

SECONDARY OUTCOMES:
Assess the psychosocial and behavioral impact of a false positive screening result. | 9 Years
Assess provider receptivity to optical spectroscopy | 9 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (4):
  - Hermann Professional Building Clinic, Houston, Texas
  - LBJ Hospital, Houston, Texas
  - Texas Medical Center Clinic, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Vancouver General Hospital/British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org